CLINICAL TRIAL: NCT03673839
Title: Randomized Clinical Trial in Healthy Men Evaluating the Impact of Dairy and Plant-based Protein Blends on Plasma Amino Acids
Brief Title: Comparison of Plant and Animal Proteins on Amino Acid Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone North America (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NU382
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Healthy Resistance-Trained Males
MeSH Terms: interventions — Crossing Over, Genetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Animal proteins (crossover) (Active Comparator)
  Interventions: Other: Animal Proteins (crossover); Other: Plant-based protein blends type 1 (crossover); Other: Plant-based protein blends type 2 (crossover); Other: Plant-based protein blends type 3 (crossover)
- Plant-based protein blends type 1 (crossover) (Experimental)
  Interventions: Other: Animal Proteins (crossover); Other: Plant-based protein blends type 1 (crossover); Other: Plant-based protein blends type 2 (crossover); Other: Plant-based protein blends type 3 (crossover)
- Plant-based protein blends type 2 (crossover) (Experimental)
  Interventions: Other: Animal Proteins (crossover); Other: Plant-based protein blends type 1 (crossover); Other: Plant-based protein blends type 2 (crossover); Other: Plant-based protein blends type 3 (crossover)
- Plant-based protein blends type 3 (crossover) (Experimental)
  Interventions: Other: Animal Proteins (crossover); Other: Plant-based protein blends type 1 (crossover); Other: Plant-based protein blends type 2 (crossover); Other: Plant-based protein blends type 3 (crossover)

INTERVENTIONS:
Other: Animal Proteins (crossover) — Animal proteins mixed with water and consumed as a beverage once by the subject in a 4x4 Williams square crossover design
Other: Plant-based protein blends type 1 (crossover) — Plant-based protein blends mixed with water and consumed as a beverage once by the subject in a 4x4 Williams square crossover design
Other: Plant-based protein blends type 2 (crossover) — Plant-based protein blends mixed with water and consumed as a beverage once by the subject in a 4x4 Williams square crossover design
Other: Plant-based protein blends type 3 (crossover) — Plant-based protein blends mixed with water and consumed as a beverage once by the subject in a 4x4 Williams square crossover design

SUMMARY:
The study purpose is to assess various protein blends, which differ in protein quality, and the impact on blood amino acid response in male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, resistance-trained adult men 18-35 years of age, inclusive, at the screening visit.
* BMI between 18.5 and 29.9 kg/m² inclusive at sceening
* Self-reported resistance training experience of no less than two years , and have participated in resistance training of at least 1h two days per week for the past six months.
* Willing to abstain from any protein supplements for 1 day prior to the study intervention phase (i.e. from the randomised visit, Visit 2)

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male subjects.
Enrollment: 20 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Plasma essential amino acids amounts | 4 hours
  Following an overnight fast, blood amino acids will be measured over 4 hours

SECONDARY OUTCOMES:
Kinetic response of the branch chain amino acids | 4 hours
  Following an overnight fast, plasma branch chain amino acids amounts (area under the curve) will be measured over 4 hours at fasting
Maximum amount of plasma branch chain amino acid amounts | 4 hours
  The maximum plasma branch chain amino acid amount will be measured over 4 hours

OTHER OUTCOMES:
Time to reach the maximum amount of plasma branch chain amino acid amounts | 4 hours
  The time to reach the maximum of plasma branch chain amino acid amount will be measured over 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jessica BRENNAN, Study Chair — Danone North America
Locations (1):
- Glycemic, Index Laboratories, Inc., Toronto, Ontario, Canada